CLINICAL TRIAL: NCT00960544
Title: Correlation of Genomic Variation in Enzymes Responsible for Metabolism of Capecitabine With Drug Metabolism Using a Limited Pharmacokinetic Sampling Plan
Brief Title: Correlation of Genomic Variation in Enzymes Responsible for Metabolism of Capecitabine With Drug Metabolism
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator departed from institution
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0003
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: Capecitabine; Xeloda; Gene expression; Pharmacokinetic testing; PK sampling; DNA analysis
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Capecitabine (Experimental): Capecitabine - Routine administration of twice daily dosing for days 1-14 of a 21-day cycle.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Routine administration of twice daily dosing for days 1-14 of a 21-day cycle.
  Other Names: Xeloda

SUMMARY:
The goal of this clinical research study is to find out how gene expression (as well as how often this expression occurs) in patients with breast cancer affects how Xeloda® (capecitabine) is cleared (passed through the urine) from the body. The safety of capecitabine will also be studied.

DETAILED DESCRIPTION:
Capecitabine, PK Testing, and DNA Analysis:

Capecitabine is designed to interfere with the growth of cancer cells, which may cause the cells to die. It is cleared from the body by certain proteins (which are made from DNA--the gene material of cells). Some patients have changes in these proteins that increase or decrease the rate that capecitabine is cleared from the body.

Researchers will use pharmacokinetic (PK) testing and DNA analysis to learn how capecitabine is cleared from your body. PK testing measures the amount of drug in the body at different time points. Information learned in this study may help researchers decide the best doses of capecitabine for future patients with breast cancer.

Screening Visit:

Before you can start treatment on this study, you will have about 2 teaspoons of blood drawn for routine tests and to make sure that you are able to receive chemotherapy. This screening blood test will help the study doctor decide if you are eligible to take part in this study.

Capecitabine Treatment:

If you are found to be eligible to take part in this study, you will be given capecitabine by mouth on the day you choose to start this therapy. Your treating doctor will prescribe capecitabine at a dose that is appropriate to treat the cancer. You can choose the start date, excluding weekends, but will need to begin therapy in the morning of the day you choose. You will have treatment with capecitabine even if you do not participate on this study.

PK Testing and DNA Analysis:

You will have blood drawn (about 2 teaspoons each time) for PK testing and DNA analysis of capecitabine at certain times throughout this study.

* For PK testing, blood will be drawn before your first dose of capecitabine, at 30, 60, and 90 minutes after the first dose, and then at 2, 6, 8, and 10 hours after the first dose.
* For DNA analysis, blood will only be drawn before you receive the first dose of capecitabine.

If your dose changes, these PK blood tests may need to be repeated.

Length of Study:

You will remain on this study for up to 6 months, unless the disease gets worse, you experience any intolerable side effects, or you decide to stop treatment with capecitabine.

This is an investigational study. Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a pathologic or cytologic diagnosis of invasive carcinoma of the breast.
2. Patients must give informed consent for protocol participation.
3. Age >/= 18 years
4. Patients must have and ECOG performance status of </=2.
5. Patients must be scheduled to receive capecitabine using a BID dosing strategy administered on days 1-14 of a 21-day cycle.
6. Patients must agree to blood draws for PK/PD sampling.
7. Patients are allowed to receive cytotoxic therapy in combination with capecitabine.
8. Patients must not require concurrent radiation, or hormonal therapy while receiving protocol therapy
9. Patients must not have an active infection requiring the use of intravenous antibiotics. The use of oral antibiotics as prophylaxis is allowed.
10. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential. Both men and women should practice an effective method of birth control while receiving capecitabine.
11. Patients must have recovered to grade <1 from all acute toxicity of previous chemotherapy, radiation or hormonal therapy and have adequate hematologic and hepatic function: Granulocyte count >/= 1,500/mcL; Platelet count >/= 100,000/mcL; Bilirubin </= 1.5 x ULN; AST and/or ALT </= 2 x ULN; Alkaline phosphatase (liver component, if fractionated) </= 2 x ULN; Serum creatinine within normal limits.

Exclusion Criteria:

1. Untreated or uncontrolled brain metastasis
2. History of prior therapy with capecitabine
3. Patient inability to take or absorb oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between genomic variation and capecitabine metabolism (measured by limited PK sampling) | PK testing blood draw before first dose of capecitabine, and at 30, 60, and 90 minutes, then 2, 6, 8, and 10 hours after first dose.
  Relationship between genomic variation and capecitabine metabolism (measured by limited PK sampling)

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Khanh Morrow, MD, Study Chair — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org